CLINICAL TRIAL: NCT04380064
Title: Internal Limiting Membrane Peeling in Proliferative Diabetic Retinopathy Patients Undergoing Vitrectomy for Tractional Retinal Detachment: a Randomized Clinical Trial
Brief Title: Internal Limiting Membrane Peeling in Proliferative Diabetic Retinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rush Eye Associates (Other)
Responsible Party: Principal Investigator, Sloan W. Rush, MD, Physician, Rush Eye Associates
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Retina 4
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Diabetic Retinopathy Visually Threatening

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Subjects undergo internal limiting membrane (ILM) peeling during vitrectomy for the indication of tractional retinal detachment
  Interventions: Procedure: ILM Peeling
- Control Group (Active Comparator): Subjects do not undergo ILM peeling during vitrectomy for the indication of tractional retinal detachment
  Interventions: Procedure: No ILM Peeling

INTERVENTIONS:
Procedure: ILM Peeling — ILM peeling performed during primary PPV for PDR
  Arms: Study Group
Procedure: No ILM Peeling — ILM peeling not performed during primary PPV for PDR
  Arms: Control Group

SUMMARY:
Subject/Participant Groups:

Study Group: Subjects undergo internal limiting membrane (ILM) peeling during vitrectomy for the indication of tractional retinal detachment Control Group: Subjects do not undergo ILM peeling during vitrectomy for the indication of tractional retinal detachment

DETAILED DESCRIPTION:
Hypothesis:

Subjects undergoing ILM peeling during vitrectomy will have lower central macular thickness on OCT, fewer postoperative epiretinal membranes, and thereby better final visual acuity to control subjects Randomization: Subjects will be randomized according to a coin toss during PPV, once Grade 2 or Grade 3 vitreoretinal adhesion has been determined: heads undergo ILM peeling, while tails do not.

Number of Subjects: With study power of 80%, a significance level of 0.05, a sample size of 60 patients for each group was calculated.

ELIGIBILITY:
Inclusion:

1. Subject age is 18-85 years.
2. Subject consents to study participation and is capable of 6 months of follow-up.
3. The subject has type I or II Diabetes Mellitus with active PDR in the study eye.
4. Best-corrected spectacle visual acuity (BCSVA) on the Snellen eye chart ranges from 20/40 to hand motions in the study eye.
5. The subject is determined to need a PPV for the indication of TRD (Grades 2 and 3).

Exclusion:

1. Subject is known to have a significant retinal/optic nerve disease otherwise unrelated to Diabetes Mellitus, which in the opinion of the examiner is responsible for two or more lines of reduced BCSVA (macular degeneration, optic neuritis, glaucoma, amblyopia, etc.) in the study eye.
2. Subject is known to have macular ischemia, which in the opinion of the examiner, is responsible for two or more lines of reduced BCSVA in the study eye.
3. Subject has a significant corneal or cataract opacity, which in the opinion of the examiner, is responsible for two or more lines of reduced BCSVA (corneal scar, ectasia, etc.) in the study eye.
4. Subject has had a previous vitrectomy (anterior or PPV) in the study eye.
5. Subject has uncontrolled neovascular glaucoma (intraocular pressure > 30 mmHg despite medical/surgical treatment) in the study eye.
6. Subject has uncontrolled hypertension (systolic > 200 mmHg or diastolic > 120 mmHg) despite adherence to a multiple anti-hypertensive medication regimen.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative ERM Development | 6 months
  Postoperative Epiretinal Membrane Development

SECONDARY OUTCOMES:
Visual Acuity | 6 months
  Rate of subjects achieving 20/50 or better Snellen visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Sloan Rush, MD, Study Chair — panhandle eye group
Locations (1):
- Hospital La Carlota, Montemorelos, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No